CLINICAL TRIAL: NCT03485690
Title: Time-based Register and Analysis of COPD Endpoints
Acronym: TRACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Gebro Pharma GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TRACE
Record Dates: First submitted 2018-02-12; First posted 2018-04-02 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: COPD
Keywords: COPD; Cohort study; Prospective
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD: COPD patients with no restrictions. The study protocol does not consider ad-hoc different patient groups. Prospective follow-up will be equally done in all recruited patients

SUMMARY:
The Time-based Register and Analysis of COPD Endpoints (TRACE) study is prospective cohort study aiming at evaluating COPD patients using simple basic tools normally used in the clinic at hand of any physician. The objective of the study is to accomplish specific aims. 1) describing the disease variation over time. 2) defining different disease behaviours; and 3) evaluating the impact of different therapeutic approaches on this behaviour in the different patient types. TRACE is a single center non-interventional prospective observational cohort study of COPD patients. Upon identification of cases, patients are followed-up in yearly visits sine die until death or lost to follow-up. Starting in 2012, during the yearly visits clinical, functional, radiological and analytical information is recorded via a standardized questionnaire. Variables recorded were: socio-demographics, tobacco history, comorbidities, clinical presentation during the previous year, exacerbations and hospitalization in the previous year, current pharmacological and non-pharmacological treatments, and complementary tests, including at least chest radiology, pre- and post-bronchodilator spirometry, and analytical results. Endpoints include a variety of clinically relevant variables including disease phenotypic expression, diagnostic measures and therapeutic responses.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Diagnosed of COPD, according to the current recommendations
* Evaluated in our COPD outpatient clinic in 2012 or the following years
* With three years of follow-up at least

Exclusion Criteria:

* Do not sign informed consent.
* With other relevant comorbidity that conditions their respiratory care

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The studied population will be composed solely of COPD patients. Adult patients with a diagnosis of COPD according to current standards (7), i.e. a tobacco history > 10 pack-years and a post-bronchodilator spirometry with an expiratory volume in the first second (FEV1) / forced vital capacity (FVC) ratio < 0.7, routinely followed-up in our outpatient clinic were selected for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Survival | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits, up to ten years
  Survival

SECONDARY OUTCOMES:
dyspnea | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  dyspnea measured by mMRC scale
Number of moderate or severe exacerbations | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  Number of moderate or severe exacerbations, as defined by GOLD 2017
FEV1 annual decline | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  FEV1 annual decline
Forced expiratory flow at 25-75% of expiration (FEF25-75) | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  Forced expiratory flow at 25-75% of expiration (FEF25-75)
Peak expiratory flow (PEF) | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  Peak expiratory flow (PEF)
Peripheral blood eosinophils count | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  Peripheral blood eosinophils count
Serum Alpha1-antitrypsin | At baseline
  Serum Alpha1-antitrypsin
Total IgE | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  Total IgE
Positive bronchial colonization | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  Positive bronchial colonization
Inhaled and oral COPD-related medication use | From date of randomization until the date of death from any cause or lost to follow-up, whichever came first, assessed in yearly visits
  Inhaled and oral COPD-related medication use

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Lopez-Campos, MD, Study Chair — Hospital Universitario Virgen del Rocio
Locations (1):
- Hospital Universitario Virgen del Rocio, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrasco Hernandez L, Caballero Eraso C, Ruiz-Duque B, Abad Arranz M, Marquez Martin E, Calero Acuna C, Lopez-Campos JL. Predictors of Single Bronchodilation Treatment Response for COPD: An Observational Study with the Trace Database Cohort. J Clin Med. 2021 Apr 15;10(8):1708. doi: 10.3390/jcm10081708. PMID 33921051
- [Derived] Carrasco Hernandez L, Caballero Eraso C, Ruiz-Duque B, Abad Arranz M, Marquez Martin E, Calero Acuna C, Lopez-Campos JL. Deconstructing Phenotypes in COPD: an Analysis of the TRACE Cohort. Arch Bronconeumol. 2022 Jan;58(1):30-34. doi: 10.1016/j.arbres.2020.12.010. Epub 2021 Jan 4. English, Spanish. PMID 33546927

DOCUMENTS (2):
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT03485690/Prot_002.pdf
  • Statistical Analysis Plan (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT03485690/SAP_003.pdf